CLINICAL TRIAL: NCT06308341
Title: Combined Effects of Virtual Reality and Motor Imagery Techniques With Routine Physical Therapy on Balance, Motor Function and Activities of Daily Living in Post Stroke Patients
Brief Title: Combined Effects of Virtual Reality and Motor Imagery Techniques With Routine Physical Therapy in Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0295
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Activities of Daily Living; Stroke; Motor Control; Randomized Clinical Trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: (Virtual Reality technique + Motor Imagery technique + Routine Physical Therapy) (Other): Participants in this group will receive Virtual Reality (VR) for and Motor Imagery (MI) training with routine physical therapy for every alternate day (3 days per week) for 12 weeks. Total 45 minutes of session.
  Routine physical therapy protocol will be given for 30 minutes. VR techniques for 10-15 minutes MI techniques for 05-10 minutes
  Interventions: Other: Virtual Reality technique + Motor Imagery technique + Routine Physical Therapy
- Group B: (Virtual Reality + Routine Physical Therapy ) (Experimental): The VR system consisted of a wall-mounted display, a Nintendo Wii box, a Wii remote, and a Wii Fit board. The participants will be instructed to stand on Wii Fit board while interacting with the VR system and playing the selected games.
  Routine physical therapy protocol will be given for 30 minutes along with cycling and walking for 10-15 minutes.
  VR techniques for 10-15 minutes.
  Interventions: Other: Virtual Reality + Routine Physical Therapy
- Group C: (Motor Imagery +Routine Physical Therapy) (Experimental): During the presentation of a video clip, patients will watch the video and afterwards try to do movement as same as shown in video.
  Routine physical therapy protocol will be given for 30 minutes along with Cycling and walking for 10-15 minutes MI techniques for 10-15 minutes
  Interventions: Other: Motor Imagery +Routine Physical Therapy

INTERVENTIONS:
Other: Virtual Reality technique + Motor Imagery technique + Routine Physical Therapy — Routine physical therapy for 30 minutes is explained as: warm up for 10 mins, stretching of lower limb and upper limb for 10 min, task specific training, gait training and balance training exercises for 15min, strengthening exercises for 10 min
  Arms: Group A: (Virtual Reality technique + Motor Imagery technique + Routine Physical Therapy)
Other: Virtual Reality + Routine Physical Therapy — Routine physical therapy protocol will be given for 30 minutes along with cycling and walking for 10-15 minutes.
  VR techniques for 10-15 minutes The first eight weeks focus on simple activities to enhance balance and motor function, such as tennis, boxing, bowling, kicking, soccer, table tilt, penguin slide, tilt city, single-leg extension, and torso twist. Exercise difficulty is adjusted based on performance, gradually progressing from easier to more challenging activities.
  Arms: Group B: (Virtual Reality + Routine Physical Therapy )
Other: Motor Imagery +Routine Physical Therapy — Routine physical therapy protocol will be given for 30 minutes along with Cycling and walking for 10-15 minutes MI techniques for 10-15 minutes The motor imagery program me will be performed in three steps; STEP I: The patients will watch the videos recorded by the examiner. STEP II: The patients will be asked to close their eyes, focus, and imagine how they are doing the task they had previously observed ten times.
  Step III: The patient will be asked to attempt the activity with his affected limbs according to the verbal command of the examiner Routine physical therapy for 30 minutes is explained as: warm up for 10 mins, stretching of lower limb and upper limb for 10 min, task specific training, gait training and balance training exercises for 15min, strengthening exercises for 10 min.
  Arms: Group C: (Motor Imagery +Routine Physical Therapy)

SUMMARY:
Stroke a devastating neurological condition, causing severe neurological challenges such as balance issues, motor function and cognitive deficits among survivors and can cause disability and death. The use of Virtual Reality and Motor Imagery in rehabilitation of neurologic disorders is on the rise. In stroke patients, VR and MI combination has not been studied. This study aims to investigate the combined effects of Virtual Reality and Motor Imagery Techniques with Routine Physical Therapy in patients with post stroke patients.

DETAILED DESCRIPTION:
This randomized control trial will be conducted at Safi Hospital Faisalabad in 7 months after the approval of synopsis, involving a sample size of 75 participants selected through convenience sampling based on the inclusion criteria. Participants will be randomly assigned to three groups using lottery method, in which Group A, will receive Virtual Reality and Motor Imagery training in conjunction with routine physical therapy three days a week for 12 weeks. Group B will receive VR and routine physical therapy, supplemented by 10-15 minutes of cycling and walking and Group C will receive routine physical therapy with MI techniques, along with 10-15 minutes of cycling and walking.

Fugal-Meyer Scale will be used to motor function, Berg Balance Scale for balance and Barthel Index will be used to assess activities of daily living. Assessment will be carried out at baseline, 6th week, 8th week and at 12th week and at 16th week after the discontinuation of treatment. The data will be entered and analyzed by using SPSS 26

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stroke of any etiology
2. Age between 40 to 65 years
3. Both genders
4. At least 6 months post-stroke onset
5. Able to follow and understand visual and verbal commands.
6. Hemiparetic
7. No prior experience with VR-based rehabilitation.
8. Able to walk with the use of walking aids or assistive devices.
9. Mini-Mental State Examination (MMSE) score equal to or greater than 24

Exclusion Criteria:

1. Presence of aphasia, apraxia, and hemineglect
2. Serious cardiovascular disease (heart failure, arrhythmias, angina pectoris or myocardial infarction)
3. Cerebellar lesion
4. Multiple brain accidents
5. Muscular disorder effect upper and lower extremities
6. History of seizures or epilepsy.
7. Patients whose injury occurred fewer than 6 months previously, considering the expected time for spontaneous recovery;
8. Patients with associated disorders such as epilepsy, and sensory and perceptual deficits such as hemineglect and Pusher syndrome;
9. Patients with osteo degenerative disorders that would prevent participation in the games or that could influence the body balance; and individuals who had cognitive and communication disorders, affecting understanding, that could compromise performance in the games
10. Inability to commit to the study schedule or attend the required therapy sessions

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 16 weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Fugal-Meyer Scale | 16 weeks
  Motor Function will be measured with Fugal-Meyer Scale. Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
Barthel Index | 16 weeks
  Activities of Daily Living will be measured with Barthel Index. The Barthel Index for Activities of Daily Living is an ordinal scale which measures a person's ability to complete activities of daily living (ADL). A score of 95 or 100 (the Barthel Index was measured in 5-point increments between 0 and 100) was considered a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reznik ME, Drake J, Margolis SA, Moody S, Murray K, Costa S, Mahta A, Wendell LC, Thompson BB, Rao SS, Barrett AM, Boukrina O, Daiello LA, Asaad WF, Furie KL, Jones RN. Deconstructing Poststroke Delirium in a Prospective Cohort of Patients With Intracerebral Hemorrhage. Crit Care Med. 2020 Jan;48(1):111-118. doi: 10.1097/CCM.0000000000004031. PMID 31567406
- [Background] Yin XJ, Wang YJ, Ding XD, Shi TM. Effects of motor imagery training on lower limb motor function of patients with chronic stroke: A pilot single-blind randomized controlled trial. Int J Nurs Pract. 2022 Jun;28(3):e12933. doi: 10.1111/ijn.12933. Epub 2021 Apr 10. PMID 33837986
- [Background] Anwar N, Karimi H, Ahmad A, Gilani SA, Khalid K, Aslam AS, Hanif A. Virtual Reality Training Using Nintendo Wii Games for Patients With Stroke: Randomized Controlled Trial. JMIR Serious Games. 2022 Jun 13;10(2):e29830. doi: 10.2196/29830. PMID 35699989
- [Background] Wang X, Carcel C, Woodward M, Schutte AE. Blood Pressure and Stroke: A Review of Sex- and Ethnic/Racial-Specific Attributes to the Epidemiology, Pathophysiology, and Management of Raised Blood Pressure. Stroke. 2022 Apr;53(4):1114-1133. doi: 10.1161/STROKEAHA.121.035852. Epub 2022 Mar 28. PMID 35344416
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Gaughan TCLS, Boe SG. Investigating the dose-response relationship between motor imagery and motor recovery of upper-limb impairment and function in chronic stroke: A scoping review. J Neuropsychol. 2022 Mar;16(1):54-74. doi: 10.1111/jnp.12261. Epub 2021 Aug 16. PMID 34396708
- [Background] Schuster-Amft C, Eng K, Suica Z, Thaler I, Signer S, Lehmann I, Schmid L, McCaskey MA, Hawkins M, Verra ML, Kiper D. Effect of a four-week virtual reality-based training versus conventional therapy on upper limb motor function after stroke: A multicenter parallel group randomized trial. PLoS One. 2018 Oct 24;13(10):e0204455. doi: 10.1371/journal.pone.0204455. eCollection 2018. PMID 30356229
- [Background] Dickstein R, Deutsch JE, Yoeli Y, Kafri M, Falash F, Dunsky A, Eshet A, Alexander N. Effects of integrated motor imagery practice on gait of individuals with chronic stroke: a half-crossover randomized study. Arch Phys Med Rehabil. 2013 Nov;94(11):2119-25. doi: 10.1016/j.apmr.2013.06.031. Epub 2013 Jul 18. PMID 23872048
- [Background] Patsaki I, Dimitriadi N, Despoti A, Tzoumi D, Leventakis N, Roussou G, Papathanasiou A, Nanas S, Karatzanos E. The effectiveness of immersive virtual reality in physical recovery of stroke patients: A systematic review. Front Syst Neurosci. 2022 Sep 22;16:880447. doi: 10.3389/fnsys.2022.880447. eCollection 2022. PMID 36211591
- [Background] Sip P, Kozlowska M, Czysz D, Daroszewski P, Lisinski P. Perspectives of Motor Functional Upper Extremity Recovery with the Use of Immersive Virtual Reality in Stroke Patients. Sensors (Basel). 2023 Jan 8;23(2):712. doi: 10.3390/s23020712. PMID 36679511
- [Background] Chen J, Or CK, Chen T. Effectiveness of Using Virtual Reality-Supported Exercise Therapy for Upper Extremity Motor Rehabilitation in Patients With Stroke: Systematic Review and Meta-analysis of Randomized Controlled Trials. J Med Internet Res. 2022 Jun 20;24(6):e24111. doi: 10.2196/24111. PMID 35723907
- [Background] Felipe FA, de Carvalho FO, Silva ER, Santos NGL, Fontes PA, de Almeida AS, Garcao DC, Nunes PS, de Souza Araujo AA. Evaluation instruments for physical therapy using virtual reality in stroke patients: a systematic review. Physiotherapy. 2020 Mar;106:194-210. doi: 10.1016/j.physio.2019.05.005. Epub 2019 Jun 5. PMID 31542173
- [Background] Lee SY, Kim DY, Sohn MK, Lee J, Lee SG, Shin YI, Kim SY, Oh GJ, Lee YH, Lee YS, Joo MC, Lee SY, Ahn J, Chang WH, Choi JY, Kang SH, Kim IY, Han J, Kim YH. Determining the cut-off score for the Modified Barthel Index and the Modified Rankin Scale for assessment of functional independence and residual disability after stroke. PLoS One. 2020 Jan 29;15(1):e0226324. doi: 10.1371/journal.pone.0226324. eCollection 2020. PMID 31995563
- [Background] Kouvelioti V, Kellis E, Kofotolis N, Amiridis I. Reliability of Single-leg and Double-leg Balance Tests in Subjects with Anterior Cruciate Ligament Reconstruction and Controls. Res Sports Med. 2015;23(2):151-66. doi: 10.1080/15438627.2015.1005292. Epub 2015 Feb 4. PMID 25649642